CLINICAL TRIAL: NCT03582852
Title: Laparoscopic Sacrocolpexy Versus Lateral Suspension With a Mesh for the Treatment of Pelvic Organ Prolapse : a Randomized Controlled Trial
Brief Title: Laparoscopic Sacrocolpexy Versus Lateral Suspension
Acronym: SUSPENSION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-43; 2017-A02650-53 (Registry Identifier: ID RCB)
Record Dates: First submitted 2018-05-22; First posted 2018-07-11 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- promontory (Active Comparator): Laparoscopic sacrocolpopexy, which consist in fixing a mesh between vaginal anterior wall
  Interventions: Procedure: Surgical treatment of genital prolapse
- laparoscopic lateral suspension (Active Comparator): The procedure consists in spreading out bilaterally, a subperitoneal T-shaped mesh in the anterior abdominal wall
  Interventions: Procedure: Surgical treatment of genital prolapse

INTERVENTIONS:
Procedure: Surgical treatment of genital prolapse — Laparoscopy performed according to the usual technique of the participating center with pneumoperitoneum between 12 and 15 mmHg. Placement of the 5 mm trocar operator left and right iliac fossa and 5 mm pubic addition.

SUMMARY:
Surgical treatment of genital prolapse can be performed by laparoscopic surgery or by vaginal surgery, with or without using meshes. Laparoscopic sacrocolpopexy, which consist in fixing a mesh between vaginal anterior wall and the promontory is the gold standard procedure to treat anterior prolapse or of the vaginal vault. Most of studies shows a success rate of 80% of this procedure.

However, access to the promontory could be difficult in patients because of adherences or anatomical reasons. This step of the procedure also exposes to risk of ureteral or vascular injuries. Recent issues have also found spondylodiscitis cases.

The technique of laparoscopic lateral suspension with mesh was developed by Dubuisson in 1998 allows not to have to approach the promontory and avoids both the risk of vascular injury and ureteral damage of laparoscopic sacrocolpopexy. Instead of attach the mesh to the promontory, the procedure consists in spreading out bilaterally, a subperitoneal T-shaped mesh in the anterior abdominal wall. The aim of this study is to compare the clinical and functional efficiency of the lateral suspension versus laparoscopic sacrocolpopexy.

It is a prospective, randomized, monocentric study compared two groups The study hypothesis is that the lateral suspension would provide correction than the laparoscopic sacrocolpopexy.

The primary outcome is the comparison of anatomic correction rates at 1 year Success is defined as 1 year Ba et C points < -1 centimeter in POP-Q international score.

Secondary endpoints are improve of quality of life evaluated with the validated P-QOL questionnaire, and complications rates, including post-operative posterior prolapse.

Number of subjects required is 72 patients, 36 in each group having a laparoscopic sacrocolpopexy or lateral suspension.

Outcomes will be evaluated at 1 month and 1 year post-operative consultation

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years old.
* Patients who agreed to participate in the study and signed informed consent.
* Patient affiliated to a social protection system.
* Surgical indication by laparoscopy of prolapse cure symptomatic of the anterior stage and / or isolated medium.

Exclusion Criteria:

* Minor patient.
* Patient refusing to sign the consent or unable to receive the necessary information to give informed consent.
* Patient not affiliated to a social protection system.
* Presence of one or more contraindication (s) to laparoscopy
* Presence of posterior prolapse requiring surgical treatment
* Need for an associated surgical procedure.
* Major people under legal protection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2021-04-20 (Actual)

PRIMARY OUTCOMES:
Evaluate cervico-urethral hypermobility | one year
  Success is defined by two points inferior at 1 centimeter in Pelvic organs prolapse quantification (POP-Q) international score. defining a symptomatic or asymptomatic state

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Olivier ARNAUD, Director, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France